CLINICAL TRIAL: NCT01841333
Title: A Phase 2 Study of PF-04449913 for the Treatment of Acute Myeloid Leukemia Patients With High Risk of Post-Allogeneic Stem Cell Transplantation Relapse
Brief Title: PF-04449913 For Patients With Acute Myeloid Leukemia at High Risk of Relapse After Donor Stem Cell Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: The Leukemia and Lymphoma Society (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-1558.cc; NCI-2013-00824 (Other: National Cancer Institute)
Record Dates: First submitted 2013-04-23; First posted 2013-04-26 (Estimated); Results first posted 2022-01-25 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2021-12

CONDITIONS: Adult Acute Myeloid Leukemia in Remission; Recurrent Adult Acute Myeloid Leukemia
Keywords: Myeloid leukemia in remission; Recurrent myeloid leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Myeloid | interventions — glasdegib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PF-04449913 (Experimental): Beginning 80 days after allogeneic stem cell transplant, patients receive PF-04449913 (100mg) orally once daily on days 1-28. Treatment repeats every 28 days for up to 1 year in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: PF-04449913

INTERVENTIONS:
Drug: PF-04449913 — 100mg given orally
  Other Names: Hedgehog inhibitor

SUMMARY:
This phase II trial will test whether the Hedgehog signaling pathway inhibitor PF-04449913 can decrease disease relapse in high-risk patients with acute myeloid leukemia after donor stem cell transplant.

DETAILED DESCRIPTION:
Disease relapse is the most common cause of death after allogeneic stem cell transplantation for acute myeloid leukemia. Patients at high risk for relapse may benefit from a novel, biologically rational therapeutic intervention to prevent this outcome. PF-04449913 is a small molecule inhibitor of the hedgehog (Hh) pathway that inhibits the protein Smoothened (SMO). Aberrant Hh signaling may contribute to the survival and expansion of the leukemia stem cell, and inhibiting the Hh pathway can eliminate these cells. Therefore, targeting Hh may be a logical intervention in the post-transplantation setting for those with high risk of relapse. The investigators propose a phase 2 study of PF-04449913 in patients with acute myeloid leukemia who have received an allogeneic stem cell transplantation and are at high risk of relapse.

This is an open label, phase 2 study employing PF-04449913 in acute myeloid leukemia patients who received an allogeneic stem cell transplantation and are at high risk of relapse. Patients will receive consecutive 28-day cycles of PF-04449913 at 100 mg/day, beginning on post-transplantation day 80 +/- 10 days, after their routine post-transplant bone marrow biopsy. Treatment will continue for up to one year or until they experience toxicity or disease relapse. 50 patients will be required for a 90% power to detect a 20% difference in one-year relapse-free survival.

ELIGIBILITY:
Inclusion Criteria:

* WHO-confirmed AML
* Age ≥18 years
* Between days 28 and 50 post transplantation at the time of initiation of the study drug
* ECOG performance status ≤ 2 (See Appendix A: ECOG Performance Status Scale)
* Life expectancy > 2 months
* Recipient of a myeloablative or non-myeloablative allogeneic HSCT

  * Conditioning regimen to be prescribed at investigator's discretion, but will be prospectively defined as myeloablative or non-myeloablative
* Stable engraftment, as defined by absolute neutrophil count (ANC) ≥ 1000/mm3 and platelets ≥ 25,000/mm3
* In morphologic remission (< 5% marrow blasts) based on BM biopsy performed +/- 5 days of day 28 post- transplantation
* Without clinical signs of active central nervous system disease
* For non-myeloablative transplants, ≥50% CD3 donor chimerism at screening
* High risk of relapse after HSCT, defined as the presence of minimal residual disease as measured by flow cytometry in the absence of evidence of morphologic disease on a bone marrow biopsy prior to HSCT
* Adequate organ function as indicated by the following laboratory values:

  * Aspartate aminotransferase (AST), alanine aminotransferase, (ALT) ≤ 3.0 x institutional upper limit of normal (ULN)
  * Total bilirubin ≤ 2.0 x institutional ULN, unless documented Gilbert's syndrome
  * Either creatinine <1.5 x institutional upper limit of normal (ULN) or creatinine clearance >60 mL/min as calculated by institution's standard formula
* Serum/urine pregnancy test (for females of childbearing potential) that is negative within 72 hours prior to initiation of first dose of treatment (a patient is of childbearing potential if, in the opinion of the investigator, she is biologically capable of having children and is sexually active)
* Female patients of childbearing potential and sexually active males and female partners of childbearing potential must agree to use a highly effective method of contraception throughout the study and for at least 90 days after the last dose of assigned treatment.
* Subject is able to comply with study procedures and follow-up examinations.

Exclusion Criteria:

* Concomitant treatment with other anti-neoplastic agents, with the exception, when clinically indicated, of prophylaxis in the post-transplantation setting with intrathecal chemotherapy
* Use of any other experimental drug or therapy within 28 days of baseline
* Inability to swallow or absorb drug
* Active uncontrolled acute fungal, bacterial, or other infection that is unresponsive to therapy at time of study drug dosing
* Unstable angina pectoris
* New York Heart Association Class III or IV heart failure
* QTc interval (using Fridericia's correction formula, QTcF, if prolonged) >470 msec
* Active cardiac arrhythmias with rapid ventricular response (defined as heart rate greater than 100 beats/minute)
* Known HIV infection
* Grade III/IV acute GVHD
* Current use or anticipated need for food or drugs that are known moderate/strong CYP3A4 inducers (See Table 1 and section 5.9.2: Prohibited Concomitant Therapy), with the exception of azole antifungals, which are permitted.
* Any medical, psychiatric, addictive or other kind of disorder which compromises the ability of the subject to give written informed consent and/or to comply with procedures.
* Pregnant or lactating females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2013-04-29 (Actual); Primary Completion 2019-05-08 (Actual); Study Completion 2020-02-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel A Pollyea, MD, MS, Principal Investigator — University of Colorado, Denver
Locations (2):
- United States (2):
  - University of Colorado Cancer Center, Aurora, Colorado
  - Ohio State University, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Location: two tertiary care referral centers Dates of recruitment were April 2013 to May 2019
Period: Overall Study
Arm/Group | PF-04449913
Started | 31
Completed | 31
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- High Risk for Relapse Postallogeneic Stem Cell Transplant: AML and MDS patients at high risk for postallogeneic stem cell transplant relapse
Arm/Group | High Risk for Relapse Postallogeneic Stem Cell Transplant
Number analyzed (Participants) | 31
Age, Continuous [Median (Full Range); unit: years] | 58 [20 to 70]
Sex: Female, Male [Count of Participants; unit: Participants] — We collected data on patient sex
  Participants
    Female | 17
    Male | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race : White | 29
  Race : Black or African American | 1
  Race : American Indian or Alaska Native | 1

OUTCOME MEASURES:

1. Primary Outcome: Relapse-free Survival in Days
Description: Days after transplant until disease relapse or death as measured by Kaplan-Meier statistical method.
Time Frame: 1 year
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | PF-04449913
Number analyzed (Participants) | 31
days | 142 [28 to 336]

2. Secondary Outcome: Remission Duration
Description: Length of time before remission measured in days
Time Frame: Up to 5 years
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | PF-04449913
Number analyzed (Participants) | 31
days | 333 [87 to 787]

3. Secondary Outcome: Number of Patients With Adverse Events (AE) Related to Glasdegib
Description: Subjects will be evaluated for AEs at each visit with the NCI-CTCAE version 4.03 used as a guide for the grading of severity.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | PF-04449913
Number analyzed (Participants) | 31
Participants | 28

4. Secondary Outcome: Overall Survival of All Patients
Time Frame: 1 year
Measure: Number; unit: percentage of participants
Arm/Group | PF-04449913
Number analyzed (Participants) | 31
percentage of participants | 64.5

ADVERSE EVENTS:
Time Frame: AE's were collected over the 1 year subjects were on glasdegib
Arm/Group | PF-04449913
All-Cause Mortality (participants affected / at risk) | 19/31
Serious Adverse Events (participants affected / at risk) | 2/31
Other Adverse Events (participants affected / at risk) | 26/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-04449913 (N=31)
Worsening nausea, appetite changes (Gastrointestinal disorders) | 1
nausea (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-04449913 (N=31)
Cramping/Myalgias (Musculoskeletal and connective tissue disorders) | 8
Dysgeusia (Gastrointestinal disorders) | 4
Anorexia/Weight Loss (Metabolism and nutrition disorders) | 3
Nausea (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 1
arthralgia (Musculoskeletal and connective tissue disorders) | 1
lymphopenia (Blood and lymphatic system disorders) | 1
neutropenia (Blood and lymphatic system disorders) | 1
hypophosphatemia (Metabolism and nutrition disorders) | 1
hypocalcemia (Metabolism and nutrition disorders) | 1
hypoalbuminemia (Metabolism and nutrition disorders) | 1
hyperbilirubinemia (Hepatobiliary disorders) | 1
hypertriglyceridemia (Metabolism and nutrition disorders) | 1
LFT Increase (Hepatobiliary disorders) | 1
hyponatremia (Metabolism and nutrition disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-15): https://cdn.clinicaltrials.gov/large-docs/33/NCT01841333/Prot_SAP_000.pdf